CLINICAL TRIAL: NCT04983888
Title: A Single-center, Phase 2 Open-label Trial Evaluating the Efficacy and Safety of OBINUTUZUMAB in Treatment of Immunosuppression-dependent or Immunosuppression/Treatment-resistant Primary FSGS, or Contraindication/Patient Refusal to Take High Dose Corticosteroids
Brief Title: Obinutuzumab in Primary FSGS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Fernando Fervenza, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-003887
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Primary Focal Segmental Glomerulosclerosis
MeSH Terms: interventions — obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Primary Focal Segmental Glomerulosclerosis (FSGS) (Experimental): Subjects with immunosuppression-dependent or immunosuppression/treatment-resistant primary FSGS or contraindication/patient refusal to take high dose corticosteroids, will receive obinutuzumab 1 gram on day 1 and 1 gram on day 15, given intravenously and then an identical course at 6 months.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — 1g IV on day one and 1 g IV on day 15, followed by identical course at month 6

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Obinutuzumab in inducing complete or partial remission of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Biopsy proven Focal Segmental Glomerulosclerosis (FSGS) lesion
* Foot process effacement ≥ 80% on electron microscopy.
* Presence of nephrotic syndrome (proteinuria > 3.5g/24hrs and serum albumin < 3.5 g/dl) prior to initiation of immunosuppressive therapy.
* Resistant or dependent on therapy, including corticosteroids or calcineurin inhibitors or who have failed rituximab. Patient who have contraindication to or refuse to take high dose corticosteroids are allowed.

Exclusion Criteria:

* Genetic or secondary forms of FSGS.
* Hepatitis B, C or HIV positive.
* Pregnant or breast-feeding.
* Active infection.
* Kidney transplant.
* Anemia with Hgb < 8.0 g/dL.
* Thrombocytopenia with platelet count < 100'000.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complication.
* Patients who have received cyclophosphamide in the last 6 months.
* Patients who received rituximab previously with CD20 count of < 5 cells/microliter at the time of enrollment.
* For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of less than (<) 1 percent (%) per year, during the treatment period and for at least 18 months after the last dose of study drug.
* For men: agreement to remain abstinent or use two adequate methods for contraception, including at least one method with failure rate of less than 1% per year during the treatment period and for at least 6 months (180 days) after the last dose of drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Change in proteinuria | Baseline, 6 months, 12 months
  Measured using 24 hour urine collection reported in mg/24h

SECONDARY OUTCOMES:
Remission status at 6 months | 6 months
  The number of subjects to reach either complete remission or partial remission at 12 months after infusion. Complete remission defined as proteinuria < 0.3g/24 hrs. and no more than 20% decline in eGFR. Partial remission defined as 50% reduction in proteinuria and proteinuria < 3.5 g/24hrs and no more than 20% decline in eGFR.
Remission status at 12 months | 12 months
  The number of subjects to reach either complete remission or partial remission at 12 months after infusion. Complete remission defined as proteinuria < 0.3g/24 hrs. and no more than 20% decline in eGFR. Partial remission defined as 50% reduction in proteinuria and proteinuria < 3.5 g/24hrs and no more than 20% decline in eGFR.
Change in serum albumin | Baseline, 6 months, 12 months
  Blood serum collected and reported in g/dL
Serious Adverse Events (SAEs) | 24 months
  Number of subjects to experience serious adverse events including serious infection defined as severe UTI or pyelonephritis, pneumonias or other systemic infections requiring hospitalization
Proteinuria at 18 months | 18 months
  Measured using 24 hour urine collection reported in mg/24h
Proteinuria at 24 months | 24 months
  Measured using 24 hour urine collection reported in mg/24h

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fervenza, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Dossier C, Bonneric S, Baudouin V, Kwon T, Prim B, Cambier A, Couderc A, Moreau C, Deschenes G, Hogan J. Obinutuzumab in Frequently Relapsing and Steroid-Dependent Nephrotic Syndrome in Children. Clin J Am Soc Nephrol. 2023 Dec 1;18(12):1555-1562. doi: 10.2215/CJN.0000000000000288. Epub 2023 Sep 6. PMID 37678236